CLINICAL TRIAL: NCT03456960
Title: A Phase 1, Randomized, Open-Label, Crossover Study to Evaluate the Bioequivalence of Single Oral Dose of TAK-438ASA Tablet and Single Oral Dose of TAK-438 Tablet Plus Aspirin Enteric-Coated Tablet (Study 1) and the Food Effect of Single Oral Dose of TAK-438ASA Tablet (Study 2) in Healthy Adult Male Subjects
Brief Title: A Study to Evaluate the Bioequivalence (BE) and the Food Effect of TAK-438ASA Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-438ASA-1001; U1111-1208-7631 (Registry Identifier: WHO); JapicCTI-183885 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pilot phase of Study 1,TAK-438ASA + TAK-438 and Aspirin (Experimental): One TAK-438ASA tablet, orally without breakfast, on Day 1 of Period 1 in the Pilot phase of Study 1 (Day 1), followed by a washout period (Days 2 to 15), followed by one TAK-438 10 mg tablet and one aspirin 100 mg tablet, orally without breakfast, on Day 1 of Period 2 in the Pilot phase of Study 1 (Day 16).
  Interventions: Drug: TAK-438ASA; Drug: TAK-438; Drug: Aspirin
- Pilot phase of Study 1,TAK-438 and Aspirin + TAK-438ASA (Experimental): One TAK-438 10 mg tablet and one aspirin 100 mg tablet, orally without breakfast, on Day 1 of Period 1 in the Pilot phase of Study 1 (Day 1), followed by a washout period (Days 2 to 15), followed by, one TAK-438ASA tablet, orally without breakfast, on Day 1 of Period 2 in the Pilot phase of Study 1 (Day 16).
  Interventions: Drug: TAK-438ASA; Drug: TAK-438; Drug: Aspirin
- Pivotal phase of Study 1, TAK-438ASA + TAK-438 and Aspirin (Experimental): One TAK-438ASA tablet, orally without breakfast, on Day 1 of Period 1 in the Pivotal phase of Study 1 (Day 1), followed by a washout period (Days 2 to 15), followed by one TAK-438 10 mg tablet and one aspirin 100 mg tablet, orally without breakfast, on Day 1 of Period 2 in the Pivotal phase of Study 1 (Day 16).
  Interventions: Drug: TAK-438ASA; Drug: TAK-438; Drug: Aspirin
- Pivotal phase of Study 1, TAK-438 and Aspirin + TAK-438ASA (Experimental): One TAK-438 10 mg tablet and one aspirin 100 mg tablet, orally without breakfast, on Day 1 of Period 1 in the Pivotal phase of Study 1 (Day 1), followed by a washout period (Days 2 to 15), followed by one TAK-438ASA tablet, orally without breakfast, on Day 1 of Period 2 in the Pivotal phase of Study 1 (Day 16).
  Interventions: Drug: TAK-438ASA; Drug: TAK-438; Drug: Aspirin
- Study 2,TAK-438ASA (Fasted + Fed condition) (Experimental): One TAK-438ASA tablet, orally without breakfast, on Day 1 of Period 1 in Study 2 (Day 1), followed by a washout period (Days 2 to 15), followed by one TAK-438ASA tablet, orally 30 minutes after breakfast, on Day 1 of Period 2 in Study 2 (Day 16).
  Interventions: Drug: TAK-438ASA
- Study 2,TAK-438ASA (Fed + Fasted condition) (Experimental): One TAK-438ASA tablet, orally 30 minutes after breakfast, on Day 1 of Period 1 in Study 2 (Day 1), followed by a washout period (Days 2 to 15), followed by one TAK-438ASA tablet, orally without breakfast, on Day 1 of Period 2 in Study 2 (Day 16).
  Interventions: Drug: TAK-438ASA

INTERVENTIONS:
Drug: TAK-438ASA — TAK-438ASA tablet.
Drug: TAK-438 — TAK-438 tablet.
  Arms: Pilot phase of Study 1,TAK-438 and Aspirin + TAK-438ASA; Pilot phase of Study 1,TAK-438ASA + TAK-438 and Aspirin; Pivotal phase of Study 1, TAK-438 and Aspirin + TAK-438ASA; Pivotal phase of Study 1, TAK-438ASA + TAK-438 and Aspirin
Drug: Aspirin — Aspirin enteric-coated tablet.
  Arms: Pilot phase of Study 1,TAK-438 and Aspirin + TAK-438ASA; Pilot phase of Study 1,TAK-438ASA + TAK-438 and Aspirin; Pivotal phase of Study 1, TAK-438 and Aspirin + TAK-438ASA; Pivotal phase of Study 1, TAK-438ASA + TAK-438 and Aspirin

SUMMARY:
The purposes of this study are to evaluate BE between a single-dose of TAK-438ASA tablet versus a single-dose combination of TAK-438 tablet 10 milligram (mg) and aspirin enteric-coated tablet 100 mg in Japanese healthy adult men (Study 1), and to evaluate the effects of food on the pharmacokinetics of TAK-438ASA tablet in Japanese healthy adult men (Study 2).

DETAILED DESCRIPTION:
The drug under investigation in this study is called TAK-438ASA. TAK-438ASA is being tested in Japanese healthy adult men. This study consists of two studies to evaluate bioequivalence (Study 1) and the effects of food (Study 2). Study 1 (split into a Pilot phase and a Pivotal phase) will look at bioequivalence between a single-dose of TAK-438ASA tablet versus a single-dose combination of TAK-438 tablet 10 mg and aspirin enteric-coated tablet 100 mg. Study 2 will look at the effects of food on the pharmacokinetics of TAK-438ASA tablet.

The study will enroll up to 440 participants in total (Study 1 + 2). For Study 1, 12 participants per group (24 participants in total) will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups for the pilot study to estimate the sample size of Pivotal study. After pilot study, 202 participants as a maximum per group (404 participants in total) will be randomly assigned to one of the two treatment groups:

* TAK-438ASA tablet (Period 1) + TAK-438 10 mg tablet and Aspirin 100 mg tablet (Period 2)
* TAK-438 10 mg tablet and Aspirin 100 mg tablet (Period 1) + TAK-438ASA tablet (Period 2)

For Study 2, 6 participants per group (12 participants in total) will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* TAK-438ASA tablet (Fasted condition) + TAK-438ASA tablet (Fed condition)
* TAK-438ASA tablet (Fed condition) + TAK-438ASA tablet (Fasted condition) This single-center trial will be conducted in Japan. The overall time to participate in this study is approximately 18 days. Participants will make two visits to the clinic and be hospitalized for eight days in total.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or sub-investigator, participants are capable of understanding the procedures required for the study and complying with its requirements.
2. Participants sign and date an informed consent form by themselves prior to the initiation of any study procedures.
3. Japanese healthy men aged greater than or equal to (>=) 20 and less than or equal to (=<) 60, inclusive, at the time of consent.
4. Body weight >=50 kilogram (kg) as well as body mass index (BMI) >=18.5 kilogram per meter square (kg/m^2) and =<25.0 kg/m^2 at screening test.

Exclusion Criteria:

1. Participants who received study drug within 16 weeks (112 days) prior to the start of study treatment in Period 1.
2. Participants who received TAK-438 or aspirin in a previous study.
3. Staffs at the study site and their family, or participants who depend on the study-related staffs at the study site (example, husband and wife, parents, children, brothers and sisters), or participants who may be constrained to consent to the study.
4. Participants with uncontrolled and clinically significant neurological, cardiovascular, lung, hepatic, renal, metabolic, gastrointestinal, urinary or endocrine disease, or other abnormalities (except for diseases investigated) that might affect the study participation or impact the results of the study.
5. Participants with a previous or current history of aspirin asthma (asthmatic attack induced by non-steroidal anti-inflammatory drugs, etc.).
6. Participants with hypersensitivity for components of TAK-438 tablet or aspirin enteric-coated tablet, or salicylic acid-based products.
7. Positive result in urinary test for illegal drug abuse at screening.
8. Participants who have a history of illegal drug abuse or alcoholism within the past 2 years prior to the screening visit, or who are not willing to refrain from alcohol consumption and drug use during the study period.
9. Participants who ingested a medicine, a supplement or food forbidden to be used in combination during the specified time period.
10. Participants with a current history or recent episodes (within the past 6 months) of gastrointestinal diseases (malabsorption, gastroesophageal reflux, peptic ulcer disease, erosive oesophagitis), frequent (at least once per week) heartburn or surgical intervention that might affect drug absorption.
11. Participants with a history of cancer, except for basal cell carcinoma in remission for >=5 years prior to Day 1.
12. Positive results at screening for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological test for syphilis.
13. Participants who have difficulties in blood draw from peripheral veins.
14. Participants who had >=200 milliliter (mL) of whole blood drawn within 4 weeks (28 days) prior to the start of study treatment in Period 1 or who had >=400 mL of whole blood drawn within 12 weeks (84 days) prior to the start of study treatment in Period 1.
15. Participants who had a total of >=800 mL of whole blood drawn within 52 weeks (364 days) prior to the start of study treatment in Period 1.
16. Participants who had blood components drawn within 2 weeks (14 days) prior to the start of study treatment in Period 1.
17. Clinically significant abnormalities in electrocardiogram at screening or admission (Day -1).
18. Participants with abnormal laboratory parameters suggestive of clinically significant underlying diseases or who have abnormal values in the following measures at screening: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) over the upper limit of normal.
19. Participants who are unlikely to comply with the protocol or deemed ineligible due to other reasons by the principal investigator or other investigators.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 276 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 8 March 2018 to 12 October 2018.
Pre-assignment Details: Healthy male participants were enrolled in this 2-period cross-over design study to receive 1 of the 2 treatment sequences: fixed dose combination (FDC) of TAK-438 and aspirin (TAK-438ASA) or a free combination of TAK-438 and aspirin in Study 1, and to receive 1 of the 2 sequences: FDC of TAK-438ASA under fasted or fed conditions in Study 2.
Groups:
- Pilot Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin: TAK-438 10 milligram (mg) and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 14 days, further followed by TAK-438 10 mg, tablet and aspirin 100 mg, tablet (free combination), orally, under fasted condition, once on Day 1 of Period 2.
- Pilot Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA; Pivotal Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA: TAK-438 10 mg, tablet and aspirin 100 mg, tablet (free combination), orally, under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 14 days, further followed by TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fasted condition, once on Day 1 of Period 2.
- Pivotal Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin: TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 14 days, further followed by TAK-438 10 mg, tablet and aspirin 100 mg, tablet (free combination), orally, under fasted condition, once on Day 1 of Period 2.
- Study 2, Sequence C: TAK-438ASA (Fasted + Fed Condition): TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 14 days, further followed by TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fed condition, once on Day 1 of Period 2.
- Study 2, Sequence D: TAK-438ASA (Fed + Fasted Condition): TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fed condition, once on Day 1 of Period 1, followed by a washout period of at least 14 days, further followed by TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fasted condition, once on Day 1 of Period 2.
Period: Period 1 (1 Day)
Arm/Group | Pilot Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pilot Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Pivotal Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pivotal Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Study 2, Sequence C: TAK-438ASA (Fasted + Fed Condition) | Study 2, Sequence D: TAK-438ASA (Fed + Fasted Condition)
Started | 12 | 12 | 120 | 120 | 6 | 6
Completed | 12 | 12 | 120 | 120 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | Pilot Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pilot Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Pivotal Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pivotal Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Study 2, Sequence C: TAK-438ASA (Fasted + Fed Condition) | Study 2, Sequence D: TAK-438ASA (Fed + Fasted Condition)
Started | 12 | 12 | 120 | 120 | 6 | 6
Completed | 12 | 12 | 119 | 118 | 6 | 6
Not Completed | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0 | 0
Period: Period 2 (1 Day)
Arm/Group | Pilot Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pilot Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Pivotal Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pivotal Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Study 2, Sequence C: TAK-438ASA (Fasted + Fed Condition) | Study 2, Sequence D: TAK-438ASA (Fed + Fasted Condition)
Started | 12 | 12 | 119 | 118 | 6 | 6
Completed | 11 | 12 | 119 | 117 | 6 | 6
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pilot Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Pivotal Study 1, Sequence A: TAK-438ASA + TAK-438 and Aspirin | Pivotal Study 1, Sequence B: TAK-438 and Aspirin + TAK-438ASA | Study 2, Sequence C: TAK-438ASA (Fasted + Fed Condition) | Study 2, Sequence D: TAK-438ASA (Fed + Fasted Condition) | Total
Number analyzed (Participants) | 12 | 12 | 120 | 120 | 6 | 6 | 276
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 20 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 20 and 60 years | 12 | 12 | 120 | 120 | 6 | 6 | 276
  Greater than (>) 60 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 12 | 120 | 120 | 6 | 6 | 276
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 12 | 12 | 120 | 120 | 6 | 6 | 276
Consumption of caffeine [Count of Participants; unit: Participants]
  Had caffeine consumption | 6 | 5 | 23 | 18 | 2 | 1 | 55
  Had no caffeine consumption | 6 | 7 | 97 | 102 | 4 | 5 | 221
Consumption of alcohol [Count of Participants; unit: Participants]
  Drank daily | 2 | 0 | 1 | 3 | 0 | 0 | 6
  Drank a few times per week | 2 | 2 | 9 | 9 | 0 | 0 | 22
  Drank a few times per month | 3 | 5 | 72 | 68 | 3 | 3 | 154
  Never drank | 5 | 5 | 38 | 40 | 3 | 3 | 94
Smoking classification [Count of Participants; unit: Participants]
  Never smoked | 7 | 6 | 81 | 76 | 4 | 4 | 178
  Current smoker | 2 | 0 | 9 | 12 | 1 | 1 | 25
  Ex-smoker | 3 | 6 | 30 | 32 | 1 | 1 | 73

OUTCOME MEASURES:

1. Primary Outcome: Study 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Free Base of TAK-438 (TAK-438F)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The pharmacokinetic (PK) analysis set was defined as all participants who received at least one dose of study drug, who had no major protocol deviation, and whose PK data were evaluable. Samples were not collected for Pivotal Study 1 because sufficient results were available for TAK-438F from the Pilot Study 1.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Pilot Study 1: TAK-438ASA; Pivotal Study 1: TAK-438ASA: TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fasted condition, once on Day 1 of either Period 1 or 2.
- Pilot Study 1: TAK-438 and Aspirin; Pivotal Study 1: TAK-438 and Aspirin: TAK-438 10 mg, tablet and aspirin 100 mg, tablet (free combination), orally, under fasted condition, once on Day 1 of either Period 1 or 2.
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 0 | 0
hour*nanogram per milliliter (h*ng/mL) | 92.46 (32.128) | 91.95 (31.431) |  |
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — The difference in the least square means (LSM) between study medications (TAK-438ASA tablet - concomitant administration of TAK-438 tablet and aspirin enteric-coated tablet) and the two-sided 90 percent (%) confidence interval (CI) were provided using a crossover analysis of variance (ANOVA) model. The ANOVA model included a log-transformed (natural log) analysis variable as the dependent variable, and study medication, sequence, and period as independent variables; LSM Difference = 0.0059, 90% CI 2-sided [-0.0340 to 0.0458]

2. Primary Outcome: Study 1, Cmax: Maximum Observed Plasma Concentration for TAK-438F
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK analysis set was defined as all participants who received at least one dose of study drug, who had no major protocol deviation, and whose PK data were evaluable. Samples were not collected for Pivotal Study 1 because sufficient results were available for TAK-438F from the Pilot Study 1.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 0 | 0
nanogram per milliliter (ng/mL) | 13.87 (5.0945) | 13.22 (5.0778) |  |
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — The difference in the LSM between study medications (TAK-438ASA tablet - concomitant administration of TAK-438 tablet and aspirin enteric-coated tablet) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included a log-transformed (natural log) analysis variable as the dependent variable, and study medication, sequence, and period as independent variables; LSM Difference = 0.0508, 90% CI 2-sided [-0.0079 to 0.1096]

3. Primary Outcome: Study 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Unchanged Aspirin
Time Frame: Day 1 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: The PK analysis set was defined as all participants who received at least one dose of study drug, who had no major protocol deviation, and whose PK data were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 233 | 233
h*ng/mL | 873.5 (220.94) | 831.9 (350.69) | 912.3 (327.58) | 832.7 (323.46)
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — Pilot Study 1: The difference in the LSM between study medications (TAK-438ASA tablet - concomitant administration of TAK-438 tablet and aspirin enteric-coated tablet) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included a log-transformed (natural log) analysis variable as the dependent variable, and study medication, sequence, and period as independent variables; LSM Difference = 0.0546, 90% CI 2-sided [-0.0941 to 0.2034]
Statistical Analysis 2: Comparison: Pivotal Study 1: TAK-438ASA vs Pivotal Study 1: TAK-438 and Aspirin; Test type: Equivalence — Pivotal Study 1: The difference in the LSM between study medications (TAK-438ASA tablet - concomitant administration of TAK-438 tablet and aspirin enteric-coated tablet) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model will include a log-transformed (natural log) analysis variable as the dependent variable, and study medication, sequence, and period as independent variables; LSM Difference = 0.0912, 90% CI 2-sided [0.0399 to 0.1424]

4. Primary Outcome: Study 1, Cmax: Maximum Observed Plasma Concentration for Unchanged Aspirin
Time Frame: Day 1 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 233 | 233
ng/mL | 647.6 (326.77) | 597.5 (507.90) | 701.8 (349.18) | 558.0 (404.26)
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; LSM Difference = 0.0916, 90% CI 2-sided [-0.1330 to 0.3162]
Statistical Analysis 2: Comparison: Pivotal Study 1: TAK-438ASA vs Pivotal Study 1: TAK-438 and Aspirin; Test type: Equivalence — Pivotal Study 1: The difference in the LSM between study medications (TAK-438ASA tablet - concomitant administration of TAK-438 tablet and aspirin enteric-coated tablet) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included a log-transformed (natural log) analysis variable as the dependent variable, and study medication, sequence, and period as independent variables; LSM Difference = 0.2293, 90% CI 2-sided [0.1519 to 0.3068]

5. Secondary Outcome: Study 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK analysis set included all participants who received at least one dose of study drug, who had no major protocol deviation, and whose PK data were evaluable. Samples were not collected for Pivotal Study 1 because sufficient results were available for TAK-438F from the Pilot Study 1.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 0 | 0
h*ng/mL | 94.71 (32.334) | 93.78 (31.828) |  |
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; LSM Difference = 0.0100, 90% CI 2-sided [-0.0299 to 0.0500]

6. Secondary Outcome: Study 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-438F
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 0 | 0
hour | 1.500 [1.00 to 3.00] | 1.500 [1.00 to 3.00] |  |
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; LSM Difference = -0.0281, 90% CI 2-sided [-0.1662 to 0.1100]

7. Secondary Outcome: Study 1, MRT (Infinity,ev): Mean Residence Time From Time 0 to Infinity for TAK-438F
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 0 | 0
hour | 9.610 (1.2440) | 9.751 (1.3853) |  |
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; LSM Difference = -0.0150, 90% CI 2-sided [-0.0448 to 0.0149]

8. Secondary Outcome: Study 1, Lambda (z): Terminal Disposition Phase Rate Constant for TAK-438F
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1 per hour
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 0 | 0
1 per hour | 0.08565 (0.0090230) | 0.08788 (0.013025) |  |
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; LSM Difference = -0.0195, 90% CI 2-sided [-0.0676 to 0.0286]

9. Secondary Outcome: Study 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Unchanged Aspirin
Time Frame: Day 1 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: The PK analysis set was defined as all participants who received at least one dose of study drug, who had no major protocol deviation, and whose PK data were evaluable. The PK analysis set where data at specified time points was available.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 231 | 221
h*ng/mL | 876.5 (221.10) | 834.6 (349.28) | 915.8 (328.82) | 855.4 (322.27)
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; LSM Difference = 0.0547, 90% CI 2-sided [-0.0937 to 0.2032]
Statistical Analysis 2: Comparison: Pivotal Study 1: TAK-438ASA vs Pivotal Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 4, analysis 2]; LSM Difference = 0.0654, 90% CI 2-sided [0.0141 to 0.1167]

10. Secondary Outcome: Study 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Unchanged Aspirin
Time Frame: Day 1 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 233 | 233
hour | 4.000 [2.50 to 8.50] | 4.500 [3.00 to 8.50] | 4.000 [2.00 to 11.0] | 4.500 [1.00 to 12.0]
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; LSM Difference = -0.1460, 90% CI 2-sided [-0.2478 to -0.0443]
Statistical Analysis 2: Comparison: Pivotal Study 1: TAK-438ASA vs Pivotal Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 4, analysis 2]; LSM Difference = -0.1674, 90% CI 2-sided [-0.2084 to -0.1264]

11. Secondary Outcome: Study 1, MRT (Infinity,ev): Mean Residence Time From Time 0 to Infinity for Unchanged Aspirin
Time Frame: Day 1 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 231 | 221
hour | 4.629 (1.4634) | 5.194 (1.5154) | 4.398 (1.0552) | 5.152 (2.0334)
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; LSM Difference = -0.1193, 90% CI 2-sided [-0.2179 to -0.0206]
Statistical Analysis 2: Comparison: Pivotal Study 1: TAK-438ASA vs Pivotal Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 4, analysis 2]; LSM Difference = -0.1366, 90% CI 2-sided [-0.1730 to -0.1002]

12. Secondary Outcome: Study 1, Lambda (z): Terminal Disposition Phase Rate Constant for Unchanged Aspirin
Time Frame: Day 1 pre-dose and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 1 per hour
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin
Number analyzed (Participants) | 23 | 23 | 231 | 221
1 per hour | 1.734 (0.30398) | 1.703 (0.30765) | 1.754 (0.32224) | 1.795 (0.35228)
Statistical Analysis 1: Comparison: Pilot Study 1: TAK-438ASA vs Pilot Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; LSM Difference = 0.0148, 90% CI 2-sided [-0.0734 to 0.1030]
Statistical Analysis 2: Comparison: Pivotal Study 1: TAK-438ASA vs Pivotal Study 1: TAK-438 and Aspirin; Test type: Equivalence — [test comment as in outcome 4, analysis 2]; LSM Difference = -0.0020, 90% CI 2-sided [-0.0463 to 0.0424]

13. Secondary Outcome: Study 2, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F and Its Metabolites (M) (M-I, M-II, M-III and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 9
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Study 2: TAK-438ASA Fasted: TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fasted condition, once on Day 1 of either Period 1 or 2.
- Study 2: TAK-430ASA Fed: TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fed condition, once on Day 1 of either Period 1 or 2.
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-430ASA Fed
Number analyzed (Participants) | 12 | 12
h*ng/mL
  TAK-438F | 84.26 (16.890) | 104.3 (19.470)
  M-I | 290.4 (50.706) | 266.9 (44.125)
  M-II: number analyzed (Participants) | 12 | 9
  M-II | 50.77 (19.175) | 58.29 (63.088)
  M-III | 83.59 (15.202) | 80.25 (22.318)
  M-IV-Sul | 115.9 (37.933) | 97.60 (40.882)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-430ASA Fed; Test type: Equivalence — TAK-438F: The difference in the LSM between dosing condition (TAK-438ASA tablet taken in a fed [30 minutes after starting breakfast] - TAK-438ASA tablet taken in a fasted [without breakfast] condition) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included a log-transformed (natural log) analysis variable as the dependent variable, and dosing condition, sequence, and period as independent variables; LSM Difference = 0.2138, 90% CI 2-sided [0.1609 to 0.2667]

14. Secondary Outcome: Study 2, AUC(0-48): Area Under the Plasma Concentration-time Curve From Time 0 to Time 48 Hours Over the Dosing Interval for TAK-438F and Its Metabolites (M-I, M-II, M-III and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-430ASA Fed
Number analyzed (Participants) | 12 | 12
h*ng/mL
  TAK-438F | 82.89 (16.467) | 102.9 (18.851)
  M-I | 272.1 (49.341) | 251.9 (44.461)
  M-II | 30.80 (14.808) | 24.17 (12.927)
  M-III | 82.96 (14.931) | 79.69 (22.117)
  M-IV-Sul | 111.5 (38.376) | 93.20 (41.338)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-430ASA Fed; Test type: Equivalence — [test comment as in outcome 13, analysis 1]; LSM Difference = 0.2161, 90% CI 2-sided [0.1652 to 0.2671]

15. Secondary Outcome: Study 2, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-438F and Its Metabolites (M-I, M-II, M-III and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Study 2: TAK-438ASA Fed: TAK-438 10 mg and aspirin 100 mg FDC (TAK-438ASA), tablet, orally, under fed condition, once on Day 1 of either Period 1 or 2.
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
h*ng/mL
  TAK-438F | 82.23 (16.775) | 102.4 (19.138)
  M-I | 258.6 (49.384) | 239.5 (44.950)
  M-II | 26.86 (12.921) | 20.66 (10.882)
  M-III | 81.92 (15.032) | 78.69 (21.959)
  M-IV-Sul | 108.4 (36.884) | 89.48 (39.843)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 13, analysis 1]; LSM Difference = 0.2190, 90% CI 2-sided [0.1675 to 0.2706]

16. Secondary Outcome: Study 2, Cmax: Maximum Observed Plasma Concentration for TAK-438F and Its Metabolites (M-I, M-II, M-III and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
ng/mL
  TAK-438F | 12.73 (2.5465) | 18.35 (5.4137)
  M-I | 41.26 (9.0261) | 35.22 (9.6886)
  M-II | 2.820 (0.83815) | 2.131 (0.57491)
  M-III | 15.38 (2.7078) | 14.90 (2.2273)
  M-IV-Sul | 28.52 (7.8634) | 23.09 (7.4466)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 13, analysis 1]; LSM Difference = 0.3653, 90% CI 2-sided [0.2180 to 0.5126]

17. Secondary Outcome: Study 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-438F and Its Metabolites (M-I, M-II, M-III and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
hour
  TAK-438F | 1.500 [1.00 to 2.00] | 1.500 [1.00 to 3.00]
  M-I | 1.500 [1.00 to 1.50] | 1.500 [1.00 to 4.00]
  M-II | 4.000 [3.00 to 4.00] | 4.000 [4.00 to 10.0]
  M-III | 1.750 [1.00 to 2.00] | 2.000 [1.00 to 4.00]
  M-IV-Sul | 1.500 [1.00 to 3.00] | 2.000 [1.50 to 4.00]

18. Secondary Outcome: Study 2, T1/2z: Terminal Disposition Phase Half-life for TAK-438F and Its Metabolites (M-I, M-II, M-III and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
hour
  TAK-438F | 8.293 (1.1254) | 7.951 (0.82489)
  M-I | 9.653 (1.3591) | 9.153 (1.0688)
  M-II: number analyzed (Participants) | 12 | 9
  M-II | 12.92 (10.029) | 27.52 (38.721)
  M-III | 6.797 (2.1059) | 6.826 (1.5924)
  M-IV-Sul | 4.067 (1.4194) | 4.543 (1.6209)

19. Secondary Outcome: Study 2, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Unchanged Aspirin and Its Metabolite (Salicylic Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
h*ng/mL
  Unchanged aspirin | 817.9 (296.13) | 1008 (221.75)
  Salicylic acid | 20010 (5299.3) | 20290 (5048.4)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — Unchanged aspirin: The difference in the LSM between dosing condition (TAK-438ASA tablet taken in a fed [30 minutes after starting breakfast] - TAK-438ASA tablet taken in a fasted [without breakfast] condition) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included a log-transformed (natural log) analysis variable as the dependent variable, and dosing condition, sequence, and period as independent variables; LSM Difference = 0.2089, 90% CI 2-sided [-0.0061 to 0.4239]
Statistical Analysis 2: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — Salicylic acid: The difference in the LSM between dosing condition (TAK-438ASA tablet taken in a fed [30 minutes after starting breakfast] - TAK-438ASA tablet taken in a fasted [without breakfast] condition) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included a log-transformed (natural log) analysis variable as the dependent variable, and dosing condition, sequence, and period as independent variables; LSM Difference = 0.0140, 90% CI 2-sided [-0.0639 to 0.0918]

20. Secondary Outcome: Study 2, AUC(0-24): Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours Over the Dosing Interval for Unchanged Aspirin and Its Metabolite (Salicylic Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
h*ng/mL
  Unchanged aspirin | 816.7 (295.55) | 1007 (222.08)
  Salicylic acid | 20070 (5318.8) | 20340 (5119.5)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 19, analysis 1]; LSM Difference = 0.2099, 90% CI 2-sided [-0.0048 to 0.4246]
Statistical Analysis 2: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 19, analysis 2]; LSM Difference = 0.0137, 90% CI 2-sided [-0.0712 to 0.0986]

21. Secondary Outcome: Study 2, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Unchanged Aspirin and Its Metabolite (Salicylic Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
h*ng/mL
  Unchanged aspirin | 816.5 (295.68) | 1007 (222.45)
  Salicylic acid | 19370 (5108.5) | 19760 (4853.5)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 19, analysis 1]; LSM Difference = 0.2096, 90% CI 2-sided [-0.0054 to 0.4246]
Statistical Analysis 2: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 19, analysis 2]; LSM Difference = 0.0201, 90% CI 2-sided [-0.0690 to 0.1092]

22. Secondary Outcome: Study 2, Cmax: Maximum Observed Plasma Concentration for Unchanged Aspirin and Its Metabolite (Salicylic Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK analysis set included all participants who received at least one dose of study drug, who had no major protocol deviation, and whose PK data were evaluable.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
ng/mL
  Unchanged aspirin | 632.5 (286.18) | 949.0 (415.75)
  Salicylic acid | 4414 (930.76) | 5374 (1119.4)
Statistical Analysis 1: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 19, analysis 1]; LSM Difference = 0.4058, 90% CI 2-sided [0.0803 to 0.7312]
Statistical Analysis 2: Comparison: Study 2: TAK-438ASA Fasted vs Study 2: TAK-438ASA Fed; Test type: Equivalence — [test comment as in outcome 19, analysis 2]; LSM Difference = 0.1969, 90% CI 2-sided [0.1065 to 0.2873]

23. Secondary Outcome: Study 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Unchanged Aspirin and Its Metabolite (Salicylic Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
hour
  Unchanged aspirin | 4.500 [2.00 to 6.00] | 4.000 [2.50 to 7.00]
  Salicylic acid | 5.500 [3.50 to 6.50] | 4.500 [3.00 to 8.00]

24. Secondary Outcome: Study 2, T1/2z: Terminal Disposition Phase Half-life for Unchanged Aspirin and Its Metabolite (Salicylic Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
hour
  Unchanged aspirin | 0.3749 (0.042784) | 0.4373 (0.10311)
  Salicylic acid | 2.050 (0.32982) | 1.901 (0.26555)

25. Secondary Outcome: Study 2, Ae(0-48): Amount of Drug Excreted in Urine From Time 0 to 48 Hours for TAK-438F and Its Metabolites (M-I, M-II, M-III, and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
microgram (mcg)
  TAK-438F | 433.3 (63.305) | 583.1 (110.83)
  M-I | 150.1 (99.765) | 153.4 (61.628)
  M-II | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000)
  M-IV-Sul | 237.0 (56.783) | 196.8 (59.876)

26. Secondary Outcome: Study 2, Fe(0-48): Fraction of Administered Dose Excreted Into Urine From Time 0 to Time 48 Hours for TAK-438F and Its Metabolites (M-I, M-II, M-III and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
percentage of dose
  TAK-438F | 4.333 (0.63305) | 5.831 (1.1083)
  M-I | 1.499 (0.99551) | 1.529 (0.61494)
  M-II | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000)
  M-IV-Sul | 1.854 (0.44353) | 1.539 (0.46709)

27. Secondary Outcome: Study 2, CLR: Renal Clearance for TAK-438F and Its Metabolites (M-I, M-II, M-III, and M-IV-Sul)
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liter per hour (l/h)
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
liter per hour (l/h)
  TAK-438F | 5.213 (0.65760) | 5.604 (0.55389)
  M-I | 0.5577 (0.38695) | 0.6018 (0.21705)
  M-II | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000)
  M-IV-Sul | 2.148 (0.59016) | 2.126 (0.66434)

28. Secondary Outcome: Study 2, Ae(0-24): Amount of Drug Excreted in Urine From Time 0 to 24 Hours for Unchanged Aspirin and Its Metabolites (Salicylic Acid and Salicyluric Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
mcg
  Unchanged aspirin | 481.3 (173.04) | 817.3 (403.78)
  Salicylic acid | 2318 (1904.7) | 2076 (1159.4)
  Salicyluric acid | 80180 (9852.2) | 83800 (4019.7)

29. Secondary Outcome: Study 2, Fe(0-24): Fraction of Administered Dose Excreted Into Urine From Time 0 to Time 24 Hours for Unchanged Aspirin and Its Metabolites (Salicylic Acid and Salicyluric Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
percentage of dose
  Unchanged aspirin | 0.4813 (0.17304) | 0.8173 (0.40378)
  Salicylic acid | 3.025 (2.4834) | 2.708 (1.5127)
  Salicyluric acid | 74.02 (9.0984) | 77.34 (3.7218)

30. Secondary Outcome: Study 2, CLR: Renal Clearance for Unchanged Aspirin and Its Metabolites (Salicylic Acid and Salicyluric Acid)
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK analysis set was defined as all participants who received at least one dose of study drug, who had no major protocol deviation, and whose PK data were evaluable. Data for CLR of Salicyluric acid was not calculated since the plasma concentration of Salicyluric acid was not measured.
Measure: Mean (Standard Deviation); unit: l/h
Arm/Group | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
Number analyzed (Participants) | 12 | 12
l/h
  Unchanged aspirin | 0.6181 (0.28917) | 0.7818 (0.29682)
  Salicylic acid | 0.1135 (0.083534) | 0.1022 (0.055826)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events (AE) that started after the first dose of study drug and no more than 2 days after the last dose of study drug in Period 2 (Day 18)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Two participants discontinued the study due to an AE in Period 2 pre-dose and did not receive the study drug for Period 2.
Arm/Group | Pilot Study 1: TAK-438ASA | Pilot Study 1: TAK-438 and Aspirin | Pivotal Study 1: TAK-438ASA | Pivotal Study 1: TAK-438 and Aspirin | Study 2: TAK-438ASA Fasted | Study 2: TAK-438ASA Fed
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/237 | 0/239 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/237 | 0/239 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/24 | 0/23 | 8/237 | 3/239 | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot Study 1: TAK-438ASA (N=24) | Pilot Study 1: TAK-438 and Aspirin (N=23) | Pivotal Study 1: TAK-438ASA (N=237) | Pivotal Study 1: TAK-438 and Aspirin (N=239) | Study 2: TAK-438ASA Fasted (N=12) | Study 2: TAK-438ASA Fed (N=12)
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 6 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT03456960/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03456960/SAP_001.pdf